CLINICAL TRIAL: NCT03492125
Title: A Phase I/II Dose-Escalation and Expansion Study of the Selective PKC-β Inhibitor MS-553 in Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: A Study Of The Selective PKC-β Inhibitor MS- 553
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study is terminated due to major protocol revisions. A new study in CLL patients is planned.
Sponsor: MingSight Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS-553-103
Record Dates: First submitted 2018-03-24; First posted 2018-04-10 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Aggressive Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib; venetoclax; Rituximab; obinutuzumab

STUDY DESIGN:
Intervention Model Description: a limited 3+3 phase 1 dose escalation study with expansion cohorts
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Phase I Dose Escalation Cohort A1 (MS-553 Monotherapy) (Experimental): R/R CLL/SLL patients
  Interventions: Drug: MS-553
- Phase II Expansion Cohort A2 (MS-553 Monotherapy) (Experimental): R/R CLL/SLL patients
  Interventions: Drug: MS-553
- Phase II Expansion Cohort A3 (MS-553 Monotherapy) (Experimental): patients with aggressive lymphoma
  Interventions: Drug: MS-553
- Phase I Combination Dose Escalation Cohort B1 (Experimental): BTK inhibitor naïve CLL/SLL patients
  Interventions: Drug: MS-553; Drug: acalabrutinib
- Phase II Expansion Cohort B2 (Experimental): BTK inhibitor naïve CLL/SLL patients
  Interventions: Drug: MS-553; Drug: acalabrutinib
- Phase II Expansion Cohort B3 (Experimental): BTK inhibitor naïve CLL/SLL patients with certain gene mutations
  Interventions: Drug: MS-553; Drug: acalabrutinib
- Phase I Combination Dose Escalation Cohort C1 (Experimental): Bcl-2 inhibitor naïve CLL/SLL patients
  Interventions: Drug: MS-553; Drug: venetoclax; Drug: Rituximab; Drug: obinutuzumab
- Experimental: Phase II Expansion Cohort C2 (Experimental): Bcl-2 inhibitor naïve CLL/SLL patients
  Interventions: Drug: MS-553; Drug: venetoclax; Drug: Rituximab; Drug: obinutuzumab

INTERVENTIONS:
Drug: MS-553 — Oral, multiple dose levels
  Arms: Phase I Combination Dose Escalation Cohort B1; Phase I Combination Dose Escalation Cohort C1; Phase I Dose Escalation Cohort A1 (MS-553 Monotherapy)
Drug: MS-553 — Oral recommended phase 2 dose of MS-553
  Arms: Experimental: Phase II Expansion Cohort C2; Phase II Expansion Cohort A2 (MS-553 Monotherapy); Phase II Expansion Cohort A3 (MS-553 Monotherapy); Phase II Expansion Cohort B2; Phase II Expansion Cohort B3
Drug: acalabrutinib — Oral
  Arms: Phase I Combination Dose Escalation Cohort B1; Phase II Expansion Cohort B2; Phase II Expansion Cohort B3
Drug: venetoclax — Oral
  Other Names: Venclexta; Venclyxto
  Arms: Experimental: Phase II Expansion Cohort C2; Phase I Combination Dose Escalation Cohort C1
Drug: Rituximab — IV
  Other Names: Rituxan; MabThera
  Arms: Experimental: Phase II Expansion Cohort C2; Phase I Combination Dose Escalation Cohort C1
Drug: obinutuzumab — IV
  Other Names: Gazyva
  Arms: Experimental: Phase II Expansion Cohort C2; Phase I Combination Dose Escalation Cohort C1

SUMMARY:
A Phase I/II Dose-Escalation and Expansion Study Of The Selective PKC-Β Inhibitor MS-553 In Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion in the primary escalation and expansion cohort 1 in this study, patients must meet all of the following criteria:

1. Age 18 years or older
2. Diagnosis of chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL):

   1. History of histologically documented CLL or SLL that meets IWCLL diagnostic criteria according to the 2008 guidelines, and
   2. Indication for treatment as defined by the 2008 IWCLL guidelines, or the need for disease reduction prior to allogeneic transplantation

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for the primary escalation and expansion cohorts of this study:

1. Current or past transformation of CLL/SLL to prolymphocytic leukemia (PLL), non-Hodgkin lymphoma, or Hodgkin lymphoma aggressive lymphoma outlined in the inclusion criteria for the optional cohort.
2. Active and uncontrolled autoimmune cytopenia(s)
3. Any of the following prior therapies within 14 days prior to cycle 1, day 1:

   1. Major surgery
   2. Corticosteroids greater than 20 mg / day prednisone (or equivalent), unless used by inhalation or topical route, or unless necessary for premedication before iodinated contrast dye, or for autoimmune hemolytic anemia
   3. Cytotoxic chemotherapy or biologic therapy, excepting BCR pathway kinase inhibitors for which no wash out is required (but must be stopped before cycle 1 day 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University Of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Columbia University, Herbert Irving Comprehensive Cancer Center, New York, New York
  - The Ohio State University, James Comprehensive Cancer Center, Columbus, Ohio
  - MD Anderson Cancer Center, Department of Leukemia, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled between May 2018 and Oct. 2023
Pre-assignment Details: No participants were enrolled in Cohort B2, B3 or C2
Groups:
- Phase I Dose Escalation Cohort A1 (MS-553:100 mg BID): R/R CLL/SLL patients MS-553 Monotherapy: Oral
- Phase I Dose Escalation Cohort A1 (MS-553: 200 mg BID); Phase I Dose Escalation Cohort A1 (MS-553: 250 mg BID); Phase I Dose Escalation Cohort A1 (MS-553: 300 mg BID); Phase I Dose Escalation Cohort A1 (MS-553: 350 mg BID): Refractory/Relapsed CLL/SLL patients MS-553 Monotherapy: Oral
- Phase II Expansion Cohort A3 (MS-553 Monotherapy): patients with Richter's transformation or aggressive lymphoma
  MS-553: Oral recommended phase 2 dose of MS-553
- Phase I Combination Dose Escalation Cohort B1 (MS-553: 150 mg BID); Phase I Combination Dose Escalation Cohort B1 (MS: 553: 200 mg BID): BTK inhibitor naïve CLL/SLL patients MS-553: Oral acalabrutinib: Oral
- Phase I Combination Dose Escalation Cohort C1 (MS-553: 150 mg BID); Phase I Combination Dose Escalation Cohort C1 (MS-553: 200 mg BID): Bcl-2 inhibitor naïve CLL/SLL patients
  MS-553: Oral venetoclax: Oral Rituximab: IV obinutuzumab: IV
Period: DLT Evaluation Period
Arm/Group | Phase I Dose Escalation Cohort A1 (MS-553:100 mg BID) | Phase I Dose Escalation Cohort A1 (MS-553: 200 mg BID) | Phase I Dose Escalation Cohort A1 (MS-553: 250 mg BID) | Phase I Dose Escalation Cohort A1 (MS-553: 300 mg BID) | Phase I Dose Escalation Cohort A1 (MS-553: 350 mg BID) | Phase II Expansion Cohort A2 (MS-553 Monotherapy) | Phase II Expansion Cohort A3 (MS-553 Monotherapy) | Phase I Combination Dose Escalation Cohort B1 (MS-553: 150 mg BID) | Phase I Combination Dose Escalation Cohort B1 (MS: 553: 200 mg BID) | Phase I Combination Dose Escalation Cohort C1 (MS-553: 150 mg BID) | Phase I Combination Dose Escalation Cohort C1 (MS-553: 200 mg BID)
Started | 4 | 3 | 3 | 4 | 4 | 0 | 0 | 3 | 3 | 3 | 4
Completed | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 3 | 3 | 3 | 3
Not Completed | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Period: Dose Expansion Period
Arm/Group | Phase I Dose Escalation Cohort A1 (MS-553:100 mg BID) | Phase I Dose Escalation Cohort A1 (MS-553: 200 mg BID) | Phase I Dose Escalation Cohort A1 (MS-553: 250 mg BID) | Phase I Dose Escalation Cohort A1 (MS-553: 300 mg BID) | Phase I Dose Escalation Cohort A1 (MS-553: 350 mg BID) | Phase II Expansion Cohort A2 (MS-553 Monotherapy) | Phase II Expansion Cohort A3 (MS-553 Monotherapy) | Phase I Combination Dose Escalation Cohort B1 (MS-553: 150 mg BID) | Phase I Combination Dose Escalation Cohort B1 (MS: 553: 200 mg BID) | Phase I Combination Dose Escalation Cohort C1 (MS-553: 150 mg BID) | Phase I Combination Dose Escalation Cohort C1 (MS-553: 200 mg BID)
Started | 0 | 0 | 0 | 0 | 0 | 23 | 6 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 20 | 5 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated population included all participants who had received at least one dose of the study drug
Groups:
- Phase I Dose Escalation Cohort A1 (MS-553: 100 mg BID); Phase I Dose Escalation Cohort A1 (MS-553: 200 mg BID); Phase I Dose Escalation Cohort A1 (MS-553: 250 mg BID); Phase I Dose Escalation Cohort A1 (MS-553: 300 mg BID); Phase I Dose Escalation Cohort A1 (MS-553: 350 mg BID): R/R CLL/SLL patients
  MS-553 Monotherapy: Oral
- Phase I Combination Dose Escalation Cohort B1 (MS-553:200 mg BID): BTK inhibitor naïve CLL/SLL patients
  MS-553: Oral
  acalabrutinib: Oral
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Escalation Cohort A1 (MS-553: 100 mg BID) | Phase I Dose Escalation Cohort A1 (MS-553: 200 mg BID) | Phase I Dose Escalation Cohort A1 (MS-553: 250 mg BID) | Phase I Dose Escalation Cohort A1 (MS-553: 300 mg BID) | Phase I Dose Escalation Cohort A1 (MS-553: 350 mg BID) | Phase II Expansion Cohort A2 (MS-553 Monotherapy) | Phase II Expansion Cohort A3 (MS-553 Monotherapy) | Phase I Combination Dose Escalation Cohort B1 (MS-553: 150 mg BID) | Phase I Combination Dose Escalation Cohort B1 (MS-553:200 mg BID) | Phase I Combination Dose Escalation Cohort C1 (MS-553: 150 mg BID) | Phase I Combination Dose Escalation Cohort C1 (MS-553: 200 mg BID) | Total
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 4 | 23 | 6 | 3 | 3 | 3 | 4 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 1 | 0 | 2 | 2 | 1 | 0 | 1 | 2 | 12
  >=65 years | 3 | 2 | 2 | 3 | 4 | 21 | 4 | 2 | 3 | 2 | 2 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 1 | 3 | 8 | 1 | 1 | 2 | 0 | 2 | 21
  Male | 2 | 2 | 3 | 3 | 1 | 15 | 5 | 2 | 1 | 3 | 2 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 4 | 3 | 2 | 4 | 4 | 23 | 6 | 3 | 2 | 2 | 3 | 56
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 4 | 3 | 2 | 3 | 4 | 23 | 6 | 3 | 2 | 3 | 4 | 57
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 3 | 4 | 4 | 23 | 6 | 3 | 3 | 3 | 4 | 60

OUTCOME MEASURES:

1. Primary Outcome: The Incidence Rate of DLT and TEAE Requiring Study Drug Discontinuation
Description: DLT are defined as any of the following treatment-emergent events occurring during the DLT evaluation period. 1. Death 2. Hematologic toxicities: • Grade 4 neutropenia for ≥ 7 days • Grade 3 febrile neutropenia: absolute neutrophil count (ANC) 38.3°C (101°F) or a sustained temperature ≥38°C (100.4°F) for > 1 hour • Grade 4 thrombocytopenia ≥ 14 days (patients with baseline platelet count of ≥ 50 x 109 /L) • Grade 4 thrombocytopenia ≥ 28 days (patients with baseline platelet count < 50 x 10 9 /L) • ≥ Grade 3 thrombocytopenia associated with ≥ Grade 2 hemorrhage • New ≥ Grade 3 anemia requiring transfusion in a patient previously transfusion independent. 3. Nonhematologic toxicities: • Any other ≥ Grade 3 toxicity not reversed to any one of the following three conditions in 7 days with appropriate intervention: a) baseline; b) < Grade 1; or c) a status considered to be controlled by the SRC. • Any TEAE requiring >25% of doses of scheduled study drug to be withheld during the DLT period
Time Frame: Assessments for DLT and TEAE will occur during Cycle 1 (28 days) for A1 Cohort and B1 Cohort and Cycles 1-4 (up to 112 days) for C1 Cohort.
Population: DLT evaluable population (Phase 1 only) included all participants who had completed at least 75% of their planned doses during Cycle 1 or the DLT period, unless missed doses were due to adverse events.
Measure: Count of Participants; unit: Participants
Groups:
- Phase I Dose Escalation Cohort A1 (MS-553: 100mg BID); Phase I Dose Escalation Cohort A1 (MS-553: 200mg BID); Phase I Dose Escalation Cohort A1 (MS-553: 250mg BID); Phase I Dose Escalation Cohort A1 (MS-553: 300mg BID); Phase I Dose Escalation Cohort A1 (MS-553: 350mg BID): R/R CLL/SLL patients
  MS-553 Monotherapy: Oral
- Phase I Combination Dose Escalation Cohort B1 (MS-553-200 mg BID): BTK inhibitor naïve CLL/SLL patients
  MS-553: Oral
  acalabrutinib: Oral
Arm/Group | Phase I Dose Escalation Cohort A1 (MS-553: 100mg BID) | Phase I Dose Escalation Cohort A1 (MS-553: 200mg BID) | Phase I Dose Escalation Cohort A1 (MS-553: 250mg BID) | Phase I Dose Escalation Cohort A1 (MS-553: 300mg BID) | Phase I Dose Escalation Cohort A1 (MS-553: 350mg BID) | Phase I Combination Dose Escalation Cohort B1 (MS-553: 150 mg BID) | Phase I Combination Dose Escalation Cohort B1 (MS-553-200 mg BID) | Phase I Combination Dose Escalation Cohort C1 (MS-553: 150 mg BID) | Phase I Combination Dose Escalation Cohort C1 (MS-553: 200 mg BID)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 3 | 2 | 3 | 4
Participants
  Number of participants with DLT | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Number of participants with TEAE | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

2. Secondary Outcome: The ORR of MS-553 in Patients With CLL/SLL Whose Disease Relapsed After or Was Refractory to at Least One Prior Therapy
Description: This will be assessed according to the 2008 International Workshop on Chronic Lymphocytic Leukemia (IWCLL) Response Criteria with modifications for treatment-related lymphocytosis. Any patient who receives at least one cycle of study therapy is evaluable for response.
Time Frame: Evaluation of the efficacy endpoints related to response will incorporate the data from the first 9 cycles (up to 252 days) of treatment.
Population: Consisting of all patients who received at least one dose of study therapy of MS-553 and had at least one post-baseline efficacy evaluation.
Measure: Number; unit: percentage of participants
Groups:
- Cohort A1 (MS-553: 100 mg BID); Cohort A1 (MS-553: 200 mg BID); Cohort A1 (MS-553: 250 mg BID); Cohort A1 (MS-553: 300 mg BID); Cohort A1 (MS-553: 350 mg BID): Refractory/Relapsed CLL/SLL patients
  MS-553 Monotherapy: Oral
- Cohort A2 (MS-553 Monotherapy): Refractory/Relapsed CLL/SLL patients
  MS-553: Oral recommended phase 2 dose of MS-553
- Cohort A3 (MS-553 Monotherapy): patients with Richter's transformation or aggressive lymphoma MS-553: Oral recommended phase 2 dose of MS-553
- Phase I Combination Dose Escalation Cohort B1 (MS-553: 200 mg BID): BTK inhibitor naïve CLL/SLL patients
  MS-553: Oral acalabrutinib: Oral
Arm/Group | Cohort A1 (MS-553: 100 mg BID) | Cohort A1 (MS-553: 200 mg BID) | Cohort A1 (MS-553: 250 mg BID) | Cohort A1 (MS-553: 300 mg BID) | Cohort A1 (MS-553: 350 mg BID) | Cohort A2 (MS-553 Monotherapy) | Cohort A3 (MS-553 Monotherapy) | Phase I Combination Dose Escalation Cohort B1 (MS-553: 150 mg BID) | Phase I Combination Dose Escalation Cohort B1 (MS-553: 200 mg BID) | Phase I Combination Dose Escalation Cohort C1 (MS-553: 150 mg BID) | Phase I Combination Dose Escalation Cohort C1 (MS-553: 200 mg BID)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 19 | 4 | 3 | 3 | 3 | 3
percentage of participants | 0 | 33.3 | 100 | 66.7 | 33.3 | 42.10 | 25 | 100 | 66.7 | 100 | 100

ADVERSE EVENTS:
Time Frame: For the duration of the study drug treatment (up to 3 years)
Description: The Safety Population included all participants who were enrolled and received at least one dose of study drug
Arm/Group | Phase I Dose Escalation Cohort A1 (MS-553: 100 mg BID) | Phase I Dose Escalation Cohort A1 (MS-553: 200 mg BID) | Phase I Dose Escalation Cohort A1 (MS-553: 250 mg BID) | Phase I Dose Escalation Cohort A1 (MS-553: 300 mg BID) | Phase I Dose Escalation Cohort A1 (MS-553: 350 mg BID) | Phase II Expansion Cohort A2 (MS-553 Monotherapy) | Phase II Expansion Cohort A3 (MS-553 Monotherapy) | Phase I Combination Dose Escalation Cohort B1 (MS-553: 150 mg BID) | Phase I Combination Dose Escalation Cohort B1 (MS-553: 200 mg BID) | Phase I Combination Dose Escalation Cohort C1 (MS-553: 150 mg BID) | Phase I Combination Dose Escalation Cohort C1 (MS-553: 200 mg BID)
All-Cause Mortality (participants affected / at risk) | 1/4 | 2/3 | 1/3 | 2/4 | 2/4 | 6/23 | 3/6 | 0/3 | 0/3 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/4 | 3/3 | 1/3 | 3/4 | 3/4 | 15/23 | 3/6 | 1/3 | 2/3 | 2/3 | 2/4
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/3 | 4/4 | 4/4 | 23/23 | 6/6 | 3/3 | 3/3 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Escalation Cohort A1 (MS-553: 100 mg BID) (N=4) | Phase I Dose Escalation Cohort A1 (MS-553: 200 mg BID) (N=3) | Phase I Dose Escalation Cohort A1 (MS-553: 250 mg BID) (N=3) | Phase I Dose Escalation Cohort A1 (MS-553: 300 mg BID) (N=4) | Phase I Dose Escalation Cohort A1 (MS-553: 350 mg BID) (N=4) | Phase II Expansion Cohort A2 (MS-553 Monotherapy) (N=23) | Phase II Expansion Cohort A3 (MS-553 Monotherapy) (N=6) | Phase I Combination Dose Escalation Cohort B1 (MS-553: 150 mg BID) (N=3) | Phase I Combination Dose Escalation Cohort B1 (MS-553: 200 mg BID) (N=3) | Phase I Combination Dose Escalation Cohort C1 (MS-553: 150 mg BID) (N=3) | Phase I Combination Dose Escalation Cohort C1 (MS-553: 200 mg BID) (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0
Pneumonia parainfluenzae viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aortic thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arterial thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism arterial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Escalation Cohort A1 (MS-553: 100 mg BID) (N=4) | Phase I Dose Escalation Cohort A1 (MS-553: 200 mg BID) (N=3) | Phase I Dose Escalation Cohort A1 (MS-553: 250 mg BID) (N=3) | Phase I Dose Escalation Cohort A1 (MS-553: 300 mg BID) (N=4) | Phase I Dose Escalation Cohort A1 (MS-553: 350 mg BID) (N=4) | Phase II Expansion Cohort A2 (MS-553 Monotherapy) (N=23) | Phase II Expansion Cohort A3 (MS-553 Monotherapy) (N=6) | Phase I Combination Dose Escalation Cohort B1 (MS-553: 150 mg BID) (N=3) | Phase I Combination Dose Escalation Cohort B1 (MS-553: 200 mg BID) (N=3) | Phase I Combination Dose Escalation Cohort C1 (MS-553: 150 mg BID) (N=3) | Phase I Combination Dose Escalation Cohort C1 (MS-553: 200 mg BID) (N=4)
Anaemias NEC (Blood and lymphatic system disorders) | 4 | 3 | 0 | 0 | 3 | 5 | 0 | 0 | 2 | 0 | 1
Bleeding tendencies (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eosinophilic disorders (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytoses NEC (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Lymphatic system disorders NEC (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Neutropenias (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Thrombocytopenias (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Aortic valvular disorders (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac conduction disorders (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Cardiac signs and symptoms NEC (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pericardial disorders NEC (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Supraventricular arrhythmias (Cardiac disorders) | 3 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Ear disorders NEC (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
External ear disorders NEC (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Choroid and vitreous structural change, deposit and degeneration (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation disorders (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ocular bleeding and vascular disorders NEC (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ocular disorders NEC (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ocular sensation disorders (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1
Pupil disorders (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual disorders NEC (Eye disorders) | 0 | 1 | 0 | 1 | 2 | 5 | 1 | 1 | 3 | 0 | 2
Colitis (excl infective) (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental and periodontal infections and inflammations (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (excl infective) (Gastrointestinal disorders) | 2 | 2 | 3 | 2 | 4 | 11 | 3 | 2 | 1 | 1 | 2
Dyspeptic signs and symptoms (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 1
Flatulence, bloating and distension (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Gastrointestinal and abdominal pains (excl oral and throat) (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2 | 6 | 0 | 0 | 0 | 1 | 3
Gastrointestinal atonic and hypomotility disorders NEC (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 1 | 2 | 0 | 0 | 1 | 1 | 1
Gastrointestinal inflammatory disorders NEC (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal signs and symptoms NEC (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0
Gastrointestinal spastic and hypermotility disorders (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids and gastrointestinal varices (excl oesophageal) (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Nausea and vomiting symptoms (Gastrointestinal disorders) | 4 | 2 | 3 | 2 | 3 | 17 | 2 | 2 | 3 | 2 | 4
Oral dryness and saliva altered (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 4 | 0 | 0 | 1 | 1 | 0
Oral soft tissue pain and paraesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peritoneal and retroperitoneal disorders (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis and ulceration (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tongue signs and symptoms (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthenic conditions (General disorders) | 2 | 1 | 3 | 2 | 3 | 11 | 1 | 2 | 2 | 2 | 3
Febrile disorders (General disorders) | 2 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Feelings and sensations NEC (General disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 1
Gait disturbances (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
General signs and symptoms NEC (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Healing abnormal NEC (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Implant and catheter site reactions (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site reactions (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mucosal findings abnormal (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema NEC (General disorders) | 1 | 2 | 2 | 0 | 1 | 4 | 0 | 1 | 0 | 1 | 3
Pain and discomfort NEC (General disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Cholecystitis and cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Allergic conditions NEC (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Immunodeficiency disorders NEC (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal and gastrointestinal infections (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Bacterial infections NEC (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Candida infections (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Clostridia infections (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dental and oral soft tissue infections (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infections (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye and eyelid infections (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Female reproductive tract infections (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes viral infections (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Infections NEC (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract and lung infections (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Skin structures and soft tissue infections (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infections (Infections and infestations) | 3 | 2 | 1 | 0 | 2 | 5 | 0 | 2 | 1 | 1 | 0
Urinary tract infections (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Viral infections NEC (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Non-site specific injuries NEC (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 1 | 1 | 4 | 1 | 0 | 2 | 1 | 0
Non-site specific procedural complications (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Overdoses NEC (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Radiation injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Site specific injuries NEC (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin injuries NEC (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 5 | 2 | 0 | 1 | 0 | 2
Spinal fractures and dislocations (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burns (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaccination related complications (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Carbohydrate tolerance analyses (incl diabetes) (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coagulation and bleeding analyses (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ECG investigations (Investigations) | 0 | 1 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Liver function analyses (Investigations) | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 2
Mineral and electrolyte analyses (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Physical examination procedures and organ system status (Investigations) | 1 | 2 | 1 | 1 | 2 | 5 | 0 | 0 | 0 | 0 | 1
Platelet analyses (Investigations) | 4 | 2 | 2 | 2 | 2 | 4 | 1 | 0 | 1 | 0 | 2
Renal function analyses (Investigations) | 2 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Skeletal and cardiac muscle analyses (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tissue enzyme analyses NEC (Investigations) | 2 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 2
White blood cell analyses (Investigations) | 4 | 2 | 2 | 1 | 4 | 6 | 1 | 0 | 1 | 0 | 2
Appetite disorders (Metabolism and nutrition disorders) | 1 | 2 | 2 | 1 | 2 | 9 | 2 | 0 | 1 | 1 | 0
Calcium metabolism disorders (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 1
Disorders of purine metabolism (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrolyte imbalance NEC (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
General nutritional disorders NEC (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemic conditions NEC (Metabolism and nutrition disorders) | 4 | 2 | 1 | 0 | 3 | 2 | 0 | 1 | 1 | 0 | 1
Hypoglycaemic conditions NEC (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Magnesium metabolism disorders (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1
Metabolic alkaloses (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Phosphorus metabolism disorders (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Potassium imbalance (Metabolism and nutrition disorders) | 3 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 1
Protein metabolism disorders NEC (Metabolism and nutrition disorders) | 4 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 0
Sodium imbalance (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 0 | 1
Total fluid volume decreased (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 0
Total fluid volume increased (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Water soluble vitamin deficiencies (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthropathies NEC (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bone disorders NEC (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bone related signs and symptoms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bursal disorders (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint related signs and symptoms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Muscle pains (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Muscle related signs and symptoms NEC (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Muscle weakness conditions (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue conditions NEC (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal and connective tissue pain and discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 4 | 1 | 0 | 0 | 1 | 1
Soft tissue disorders NEC (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spine and neck deformities (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diffuse large B-cell lymphomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Endocrine neoplasms malignant and unspecified NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Skin neoplasms malignant and unspecified (excl melanoma) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Auditory nerve disorders (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Central nervous system haemorrhages and cerebrovascular accidents (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coordination and balance disturbances (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cortical dysfunction NEC (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disturbances in consciousness NEC (Nervous system disorders) | 1 | 0 | 0 | 2 | 1 | 3 | 0 | 0 | 1 | 0 | 1
Dyskinesias and movement disorders NEC (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Encephalopathies NEC (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headaches NEC (Nervous system disorders) | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 1
Lumbar spinal cord and nerve root disorders (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Memory loss (excl dementia) (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Mental impairment (excl dementia and memory loss) (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mononeuropathies (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neurological signs and symptoms NEC (Nervous system disorders) | 0 | 2 | 1 | 2 | 0 | 7 | 2 | 1 | 1 | 1 | 2
Olfactory nerve disorders (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesias and dysaesthesias (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 0 | 0 | 0 | 3
Peripheral neuropathies NEC (Nervous system disorders) | 0 | 2 | 0 | 2 | 0 | 9 | 0 | 0 | 0 | 1 | 2
Sensory abnormalities NEC (Nervous system disorders) | 0 | 2 | 0 | 1 | 1 | 3 | 0 | 0 | 1 | 2 | 1
Anxiety symptoms (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 2
Confusion and disorientation (Psychiatric disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deliria (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depressive disorders (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disturbances in initiating and maintaining sleep (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Increased physical activity levels (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep disorders NEC (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bladder and urethral symptoms (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0
Renal failure and impairment (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Urinary abnormalities (Renal and urinary disorders) | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0
Prostatic neoplasms and hypertrophy (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breathing abnormalities (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 3 | 5 | 0 | 0 | 0 | 0 | 0
Bronchial conditions NEC (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchospasm and obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conditions associated with abnormal gas exchange (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Coughing and associated symptoms (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 1 | 1 | 3 | 0 | 0 | 1 | 0 | 3
Laryngeal and adjacent sites disorders NEC (excl infections and neoplasms) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion and inflammations (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Nasal disorders NEC (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Parenchymal lung disorders NEC (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal disorders (excl infections and neoplasms) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumothorax and pleural effusions NEC (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pulmonary oedemas (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract disorders NEC (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract signs and symptoms (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1
Acnes (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecias (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Apocrine and eccrine gland disorders (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 1 | 5 | 0 | 1 | 0 | 0 | 1
Dermal and epidermal conditions NEC (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 1
Dermatitis and eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Erythemas (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Exfoliative conditions (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Nail and nail bed conditions (excl infections and infestations) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pilar disorders NEC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pruritus NEC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Purpura and related conditions (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Rashes, eruptions and exanthems NEC (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 5 | 1 | 1 | 1 | 2 | 2
Skin and subcutaneous tissue ulcerations (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin injuries and mechanical dermatoses (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin preneoplastic conditions NEC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lens therapeutic procedures (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhages NEC (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 2
Lymphoedemas (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral embolism and thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral vascular disorders NEC (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Phlebitis NEC (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vascular hypertensive disorders NEC (Vascular disorders) | 4 | 0 | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Vascular hypotensive disorders (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT03492125/Prot_SAP_001.pdf